CLINICAL TRIAL: NCT05594563
Title: TArgeting Type 1 Diabetes Using POLyamines (TADPOL): A Randomized, Double-Masked, Placebo-Controlled Phase 2 Study to Evaluate the Efficacy and Safety of Difluoromethylornithine (DFMO) to Preserve Insulin Production in Type 1 Diabetes
Brief Title: TArgeting Type 1 Diabetes Using POLyamines (TADPOL)
Acronym: TADPOL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emily K. Sims (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Cancer Prevention Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Emily K. Sims, Associate Professor of Pediatrics, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-SRA-2022-1205-M-B
Record Dates: First submitted 2022-10-12; First posted 2022-10-26 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Eflornithine

STUDY DESIGN:
Intervention Model Description: Subject are randomized to either treatment or placebo arm.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participant, Care provider and Investigator blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Active Comparator): Difluoromethylornithine (DFMO) pill ,1000mg/m2/day, for 6 months
  Interventions: Drug: DFMO
- Placebo Arm (Placebo Comparator): Placebo pill taken twice a day orally for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DFMO — DFMO orally twice a day
  Other Names: Difluoromethylornithine
  Arms: Treatment Arm
Drug: Placebo — Placebo orally twice a day
  Arms: Placebo Arm

SUMMARY:
The goal of this clinical trial is to test a drug known as DFMO in people with Type 1 Diabetes (T1D). The main question[s] it aims to answer are:

* Does it reduce stress on the cells that make insulin?
* Does it preserve what is left of the body's insulin production? Participants will take either DFMO or a placebo (looks like DFMO but has no active ingredients) two times a day for about 6 months. Participants will have 6 in person visits and 1 phone visit over a period of 12 months. Visits will include blood draws urine collection and other tests.

DETAILED DESCRIPTION:
This study will be a multicenter, double-blind, placebo-controlled, 2:1 random assigned, phase II clinical trial for individuals with recent onset type 1 diabetes. The investigators are conducting a double masked placebo-controlled intention to treat study enrolling persons with new onset T1D with documented continued residual C-peptide production. Within 45 days of screening and a run-in period during which eligibility will be determined and glycemic control optimized, subjects will have a 6-month double-masked treatment period with either DFMO or placebo. After a 6-month wash-out period the durability of effect will be assessed. Subjects will be randomly assigned either 1000mg/m2/day oral DFMO or placebo treatment at a 2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 4- ≥40 years of age with a clinical diagnosis of T1D
2. T1D clinical diagnosis with insulin start date no more than 100 days prior to the time of randomization
3. Random non-fasting C-peptide level of >0.2 pmol/mL (equivalent to >0.6ng/ml) at screening.
4. Positive for any one of the following diabetes-related autoantibodies (IAA, GAA, IA-2, or ZnT8)
5. Treatment naïve of any immunomodulatory agent
6. Normal hearing at screening, defined as acceptable results of pure-tone audiometry (<20 decibel [dB] baseline thresholds forall frequencies tested

Exclusion Criteria:

1. Presence of severe, active disease that interferes with dietary intake or requires the use of chronic medication, with the exception of well-controlled hypothyroidism and mild asthma not requiring oral steroids. Presence of any psychiatric disorder that will affect ability to participate in study.
2. Diabetes other than T1D
3. Chronic illness known to affect glucose metabolism (e.g. Cushing syndrome, polycystic ovarian disorder, cystic fibrosis) or taking medications that affect glucose metabolism (e.g. steroids, metformin)
4. Inability to swallow pills
5. Psychiatric impairment or current use of anti-psychotic medication
6. Any condition that, in the investigator's opinion, may compromise study participation or may confound the interpretation of the study results.
7. Neutropenia (< 1,500 neutrophils/μL)
8. Leukopenia (< 3,000 leukocytes /μL)
9. Lymphopenia ( < 800 lymphocytes/μL)
10. Thrombocytopenia (<100,000 platelets/μL)
11. Clinically significant anemia or Hemoglobin as defined below:

    In Adults: Hgb <12.0g/dL in females and <13.0g/dL in males In Children: 12- <18: <11.4 g/dL in females and <12.4 g/dL in males In Children: 4- <12: Hgb <11.2 g/dL
12. Impaired renal function (assessed by history and BUN/Creatinine, DFMO is renally excreted)
13. Allergy to milk or soy (components of Boost® drink used for mixed meal tolerance testing)
14. Female participants of child-bearing age with reproductive potential, must not be pregnant and agree to use 2 effective forms of birth control or be abstinent during the study period (see below). Male participants (including men who have had vasectomies) whose partners are pregnant or may be pregnant should use condoms while on study drug, until 2 weeks after discontinuation of drug, while the partner is pregnant.
15. Active seizure disorder, defined as requiring chronic medication at the time of study or having had a seizure within the past 12 months at the time of screening
16. Enrollment into another intervention trial.

Ages: 4 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy of 1000 mg/m2/day of oral DFMO after 6 months of treatment | 6 month
  Primary endpoint defining clinical efficacy will be based on mixed-meal stimulated C-peptide area under the curve (AUC; in arbitrary units) in the treatment group compared to placebo after 6 months of DFMO treatment
Number of participants with treatment-related adverse events as assessed by CTCAE v5 | through study completion, an average of one year
  A summary of serious and non-serious adverse events (AEs) will be reported.

SECONDARY OUTCOMES:
Clinical efficacy of 1000 mg/m2/day of oral DFMO after 3 months of treatment, 9 months after treatment (or 3 months after treatment end), and 12 months after treatment (or 6 months after treatment end). | through study completion, an average of one year
  Secondary endpoints will be based on mixed meal stimulated C-peptide AUC (arbitrary units) at 3 months after treatment, 9 months after treatment, and 12 months after treatment.
Decrease in urinary polyamides after 6 months of DFMO treatment. | up to 24 weeks after treatment
  Decrease in urinary putrescine (in umol/g Cr) from baseline after 6 months of DFMO treatment, measured using high performance liquid chromatography.
Biomarkers of β cell stress at 3, 6, 9, and 12 months after treatment. | through study completion, an average of one year
  Fasting and stimulated proinsulin/c-peptide ratios (%) will be measured using immunoassays and reported at baseline, 3 months after treatment, 6 months after treatment, 9 months after treatment, and 12 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Emily K Sims, MD,MS, Study Chair — Indiana University School of Medicine
Locations (7):
- United States (7):
  - Barbara Davis Center, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - IU Health Riley Hospital for Children, Indianapolis, Indiana
  - Children's Mercy Hospital, Kansas City, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - MHealth Fairview Masonic Children's Hospital and Specialty Clinics, Minneapolis, Minnesota
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooks WH. Autoimmune diseases and polyamines. Clin Rev Allergy Immunol. 2012 Feb;42(1):58-70. doi: 10.1007/s12016-011-8290-y. PMID 22116709
- [Background] Hong SK, Chaturvedi R, Piazuelo MB, Coburn LA, Williams CS, Delgado AG, Casero RA Jr, Schwartz DA, Wilson KT. Increased expression and cellular localization of spermine oxidase in ulcerative colitis and relationship to disease activity. Inflamm Bowel Dis. 2010 Sep;16(9):1557-66. doi: 10.1002/ibd.21224. PMID 20127992
- [Background] Seiler N. Catabolism of polyamines. Amino Acids. 2004 Jun;26(3):217-33. doi: 10.1007/s00726-004-0070-z. Epub 2004 Apr 20. PMID 15221502
- [Background] Jeter JM, Alberts DS. Difluoromethylornithine: the proof is in the polyamines. Cancer Prev Res (Phila). 2012 Dec;5(12):1341-4. doi: 10.1158/1940-6207.CAPR-12-0429. PMID 23221207
- [Background] Maier B, Tersey SA, Mirmira RG. Hypusine: a new target for therapeutic intervention in diabetic inflammation. Discov Med. 2010 Jul;10(50):18-23. PMID 20670594
- [Background] Maier B, Ogihara T, Trace AP, Tersey SA, Robbins RD, Chakrabarti SK, Nunemaker CS, Stull ND, Taylor CA, Thompson JE, Dondero RS, Lewis EC, Dinarello CA, Nadler JL, Mirmira RG. The unique hypusine modification of eIF5A promotes islet beta cell inflammation and dysfunction in mice. J Clin Invest. 2010 Jun;120(6):2156-70. doi: 10.1172/JCI38924. Epub 2010 May 24. PMID 20501948
- [Background] Templin AT, Maier B, Nishiki Y, Tersey SA, Mirmira RG. Deoxyhypusine synthase haploinsufficiency attenuates acute cytokine signaling. Cell Cycle. 2011 Apr 1;10(7):1043-9. doi: 10.4161/cc.10.7.15206. Epub 2011 Apr 1. PMID 21389784
- [Background] Bjelakovic G, Beninati S, Bjelakovic B, Sokolovic D, Jevtovic T, Stojanovic I, Rossi S, Tabolacci C, Kocic G, Pavlovic D, Saranac Lj, Zivic S. Does polyamine oxidase activity influence the oxidative metabolism of children who suffer of diabetes mellitus? Mol Cell Biochem. 2010 Aug;341(1-2):79-85. doi: 10.1007/s11010-010-0439-0. Epub 2010 Apr 20. PMID 20405312
- [Background] Nishiki Y, Adewola A, Hatanaka M, Templin AT, Maier B, Mirmira RG. Translational control of inducible nitric oxide synthase by p38 MAPK in islet beta-cells. Mol Endocrinol. 2013 Feb;27(2):336-49. doi: 10.1210/me.2012-1230. Epub 2012 Dec 18. PMID 23250488
- [Background] Higashi K, Yoshida M, Igarashi A, Ito K, Wada Y, Murakami S, Kobayashi D, Nakano M, Sohda M, Nakajima T, Narita I, Toida T, Kashiwagi K, Igarashi K. Intense correlation between protein-conjugated acrolein and primary Sjogren's syndrome. Clin Chim Acta. 2010 Mar;411(5-6):359-63. doi: 10.1016/j.cca.2009.11.032. Epub 2009 Dec 5. PMID 19968980
- [Background] Furumitsu Y, Yukioka K, Kojima A, Yukioka M, Shichikawa K, Ochi T, Matsui-Yuasa I, Otani S, Nishizawa Y, Morii H. Levels of urinary polyamines in patients with rheumatoid arthritis. J Rheumatol. 1993 Oct;20(10):1661-5. PMID 8295175
- [Background] Furumitsu Y, Yukioka K, Yukioka M, Ochi T, Morishima Y, Matsui-Yuasa I, Otani S, Inaba M, Nishizawa Y, Morii H. Interleukin-1beta induces elevation of spermidine/spermine N1-acetyltransferase activity and an increase in the amount of putrescine in synovial adherent cells from patients with rheumatoid arthritis. J Rheumatol. 2000 Jun;27(6):1352-7. PMID 10852253
- [Background] Bardocz S, Duguid TJ, Brown DS, Grant G, Pusztai A, White A, Ralph A. The importance of dietary polyamines in cell regeneration and growth. Br J Nutr. 1995 Jun;73(6):819-28. doi: 10.1079/bjn19950087. PMID 7632663
- [Background] Zoumas-Morse C, Rock CL, Quintana EL, Neuhouser ML, Gerner EW, Meyskens FL Jr. Development of a polyamine database for assessing dietary intake. J Am Diet Assoc. 2007 Jun;107(6):1024-7. doi: 10.1016/j.jada.2007.03.012. PMID 17524725
- [Background] Milovic V. Polyamines in the gut lumen: bioavailability and biodistribution. Eur J Gastroenterol Hepatol. 2001 Sep;13(9):1021-5. doi: 10.1097/00042737-200109000-00004. PMID 11564949
- [Background] Soda K, Kano Y, Sakuragi M, Takao K, Lefor A, Konishi F. Long-term oral polyamine intake increases blood polyamine concentrations. J Nutr Sci Vitaminol (Tokyo). 2009 Aug;55(4):361-6. doi: 10.3177/jnsv.55.361. PMID 19763038
- [Background] Sjoholm A, Arkhammar P, Berggren PO, Andersson A. Polyamines in pancreatic islets of obese-hyperglycemic (ob/ob) mice of different ages. Am J Physiol Cell Physiol. 2001 Feb;280(2):C317-23. doi: 10.1152/ajpcell.2001.280.2.C317. PMID 11208527
- [Background] Sjoholm A, Arkhammar P, Welsh N, Bokvist K, Rorsman P, Hallberg A, Nilsson T, Welsh M, Berggren PO. Enhanced stimulus-secretion coupling in polyamine-depleted rat insulinoma cells. An effect involving increased cytoplasmic Ca2+, inositol phosphate generation, and phorbol ester sensitivity. J Clin Invest. 1993 Oct;92(4):1910-7. doi: 10.1172/JCI116784. PMID 8408643
- [Background] Roy UK, Rial NS, Kachel KL, Gerner EW. Activated K-RAS increases polyamine uptake in human colon cancer cells through modulation of caveolar endocytosis. Mol Carcinog. 2008 Jul;47(7):538-53. doi: 10.1002/mc.20414. PMID 18176934
- [Background] Belting M, Mani K, Jonsson M, Cheng F, Sandgren S, Jonsson S, Ding K, Delcros JG, Fransson LA. Glypican-1 is a vehicle for polyamine uptake in mammalian cells: a pivital role for nitrosothiol-derived nitric oxide. J Biol Chem. 2003 Nov 21;278(47):47181-9. doi: 10.1074/jbc.M308325200. Epub 2003 Sep 11. PMID 12972423
- [Background] Belting M, Persson S, Fransson LA. Proteoglycan involvement in polyamine uptake. Biochem J. 1999 Mar 1;338 ( Pt 2)(Pt 2):317-23. PMID 10024506
- [Background] Welch JE, Bengtson P, Svensson K, Wittrup A, Jenniskens GJ, Ten Dam GB, Van Kuppevelt TH, Belting M. Single chain fragment anti-heparan sulfate antibody targets the polyamine transport system and attenuates polyamine-dependent cell proliferation. Int J Oncol. 2008 Apr;32(4):749-56. PMID 18360702
- [Background] Nevins AK, Thurmond DC. Caveolin-1 functions as a novel Cdc42 guanine nucleotide dissociation inhibitor in pancreatic beta-cells. J Biol Chem. 2006 Jul 14;281(28):18961-72. doi: 10.1074/jbc.M603604200. Epub 2006 May 19. PMID 16714282
- [Background] Park MH, Nishimura K, Zanelli CF, Valentini SR. Functional significance of eIF5A and its hypusine modification in eukaryotes. Amino Acids. 2010 Feb;38(2):491-500. doi: 10.1007/s00726-009-0408-7. Epub 2009 Dec 8. PMID 19997760
- [Background] Robbins RD, Tersey SA, Ogihara T, Gupta D, Farb TB, Ficorilli J, Bokvist K, Maier B, Mirmira RG. Inhibition of deoxyhypusine synthase enhances islet beta cell function and survival in the setting of endoplasmic reticulum stress and type 2 diabetes. J Biol Chem. 2010 Dec 17;285(51):39943-52. doi: 10.1074/jbc.M110.170142. Epub 2010 Oct 18. PMID 20956533
- [Background] Renaudineau Y, Youinou P. Epigenetics and autoimmunity, with special emphasis on methylation. Keio J Med. 2011;60(1):10-6. doi: 10.2302/kjm.60.10. PMID 21460598
- [Background] Packham G, Cleveland JL. The role of ornithine decarboxylase in c-Myc-induced apoptosis. Curr Top Microbiol Immunol. 1995;194:283-90. doi: 10.1007/978-3-642-79275-5_33. PMID 7895500
- [Background] Tersey SA, Nishiki Y, Templin AT, Cabrera SM, Stull ND, Colvin SC, Evans-Molina C, Rickus JL, Maier B, Mirmira RG. Islet beta-cell endoplasmic reticulum stress precedes the onset of type 1 diabetes in the nonobese diabetic mouse model. Diabetes. 2012 Apr;61(4):818-27. doi: 10.2337/db11-1293. PMID 22442300
- [Background] Watkins RA, Evans-Molina C, Terrell JK, Day KH, Guindon L, Restrepo IA, Mirmira RG, Blum JS, DiMeglio LA. Proinsulin and heat shock protein 90 as biomarkers of beta-cell stress in the early period after onset of type 1 diabetes. Transl Res. 2016 Feb;168:96-106.e1. doi: 10.1016/j.trsl.2015.08.010. Epub 2015 Sep 4. PMID 26397425
- [Background] Soda K, Kano Y, Nakamura T, Kasono K, Kawakami M, Konishi F. Spermine, a natural polyamine, suppresses LFA-1 expression on human lymphocyte. J Immunol. 2005 Jul 1;175(1):237-45. doi: 10.4049/jimmunol.175.1.237. PMID 15972654
- [Background] Hsu HC, Thomas T, Sigal LH, Thomas TJ. Polyamine-fas interactions: inhibition of polyamine biosynthesis in MRL-lpr/lpr mice is associated with the up-regulation of fas mRNA in thymocytes. Autoimmunity. 1999;29(4):299-309. doi: 10.3109/08916939908994750. PMID 10433086
- [Background] Abeloff MD, Slavik M, Luk GD, Griffin CA, Hermann J, Blanc O, Sjoerdsma A, Baylin SB. Phase I trial and pharmacokinetic studies of alpha-difluoromethylornithine--an inhibitor of polyamine biosynthesis. J Clin Oncol. 1984 Feb;2(2):124-30. doi: 10.1200/JCO.1984.2.2.124. PMID 6422008
- [Background] Pepin J, Milord F, Guern C, Schechter PJ. Difluoromethylornithine for arseno-resistant Trypanosoma brucei gambiense sleeping sickness. Lancet. 1987 Dec 19;2(8573):1431-3. doi: 10.1016/s0140-6736(87)91131-7. PMID 2891995
- [Background] Wolf JE Jr, Shander D, Huber F, Jackson J, Lin CS, Mathes BM, Schrode K; Eflornithine HCl Study Group. Randomized, double-blind clinical evaluation of the efficacy and safety of topical eflornithine HCl 13.9% cream in the treatment of women with facial hair. Int J Dermatol. 2007 Jan;46(1):94-8. doi: 10.1111/j.1365-4632.2006.03079.x. No abstract available. PMID 17214730
- [Background] Gerner EW, Meyskens FL Jr. Combination chemoprevention for colon cancer targeting polyamine synthesis and inflammation. Clin Cancer Res. 2009 Feb 1;15(3):758-61. doi: 10.1158/1078-0432.CCR-08-2235. PMID 19188144
- [Background] Lewis EC, Kraveka JM, Ferguson W, Eslin D, Brown VI, Bergendahl G, Roberts W, Wada RK, Oesterheld J, Mitchell D, Foley J, Zage P, Rawwas J, Rich M, Lorenzi E, Broglio K, Berry D, Saulnier Sholler GL. A subset analysis of a phase II trial evaluating the use of DFMO as maintenance therapy for high-risk neuroblastoma. Int J Cancer. 2020 Dec 1;147(11):3152-3159. doi: 10.1002/ijc.33044. Epub 2020 May 24. PMID 32391579
- [Background] Bowlin TL, McKown BJ, Davis GF, Sunkara PS. Effect of polyamine depletion in vivo by DL-alpha-difluoromethylornithine on functionally distinct populations of tumoricidal effector cells in normal and tumor-bearing mice. Cancer Res. 1986 Nov;46(11):5494-8. PMID 3093066
- [Background] Mari A, Tura A, Gastaldelli A, Ferrannini E. Assessing insulin secretion by modeling in multiple-meal tests: role of potentiation. Diabetes. 2002 Feb;51 Suppl 1:S221-6. doi: 10.2337/diabetes.51.2007.s221. PMID 11815483
- [Background] Gitelman SE, Bundy BN, Ferrannini E, Lim N, Blanchfield JL, DiMeglio LA, Felner EI, Gaglia JL, Gottlieb PA, Long SA, Mari A, Mirmira RG, Raskin P, Sanda S, Tsalikian E, Wentworth JM, Willi SM, Krischer JP, Bluestone JA; Gleevec Trial Study Group. Imatinib therapy for patients with recent-onset type 1 diabetes: a multicentre, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Diabetes Endocrinol. 2021 Aug;9(8):502-514. doi: 10.1016/S2213-8587(21)00139-X. Epub 2021 Jun 29. PMID 34214479
- [Background] Metcalf BW, Bey P, Danzin C, Jung MJ, Casara P, Vevert JP: Catalytic irreversible inhibition of mammalian ornithine decarboxylase (E.C.4.1.1.17) by substrate and product analogs. Journal of the American Chemical Society 1978;100:2551-2553
- [Background] Poulin R, Lu L, Ackermann B, Bey P, Pegg AE. Mechanism of the irreversible inactivation of mouse ornithine decarboxylase by alpha-difluoromethylornithine. Characterization of sequences at the inhibitor and coenzyme binding sites. J Biol Chem. 1992 Jan 5;267(1):150-8. PMID 1730582
- [Background] Pegg AE, McGovern KA, Wiest L. Decarboxylation of alpha-difluoromethylornithine by ornithine decarboxylase. Biochem J. 1987 Jan 1;241(1):305-7. doi: 10.1042/bj2410305. PMID 3105526
- [Background] Selamnia M, Mayeur C, Robert V, Blachier F. Alpha-difluoromethylornithine (DFMO) as a potent arginase activity inhibitor in human colon carcinoma cells. Biochem Pharmacol. 1998 Apr 15;55(8):1241-5. doi: 10.1016/s0006-2952(97)00572-8. PMID 9719479
- [Background] Danzin C, Jung MJ, Grove J, Bey P. Effect of alpha-difluoromethylornithine, an enzyme-activated irreversible inhibitor of ornithine decarboxylase, on polyamine levels in rat tissues. Life Sci. 1979 Feb 5;24(6):519-24. doi: 10.1016/0024-3205(79)90173-5. No abstract available. PMID 431333
- [Background] Oredsson S, Anehus S, Heby O. Inhibition of cell proliferation by DL-alpha-difluoromethylornithine, a catalytic irreversible inhibitor of ornithine decarboxylase. Acta Chem Scand B. 1980;34(6):457-8. doi: 10.3891/acta.chem.scand.34b-0457. No abstract available. PMID 6781187
- [Background] Pena A, Reddy CD, Wu S, Hickok NJ, Reddy EP, Yumet G, Soprano DR, Soprano KJ. Regulation of human ornithine decarboxylase expression by the c-Myc.Max protein complex. J Biol Chem. 1993 Dec 25;268(36):27277-85. PMID 8262968
- [Background] Bello-Fernandez C, Packham G, Cleveland JL. The ornithine decarboxylase gene is a transcriptional target of c-Myc. Proc Natl Acad Sci U S A. 1993 Aug 15;90(16):7804-8. doi: 10.1073/pnas.90.16.7804. PMID 8356088
- [Background] Celano P, Baylin SB, Giardiello FM, Nelkin BD, Casero RA Jr. Effect of polyamine depletion on c-myc expression in human colon carcinoma cells. J Biol Chem. 1988 Apr 25;263(12):5491-4. PMID 3128541
- [Background] Tabib A, Bachrach U. Role of polyamines in mediating malignant transformation and oncogene expression. Int J Biochem Cell Biol. 1999 Nov;31(11):1289-95. doi: 10.1016/s1357-2725(99)00098-9. PMID 10605821
- [Background] Liu R, Jia Y, Cheng W, Ling J, Liu L, Bi K, Li Q. Determination of polyamines in human urine by precolumn derivatization with benzoyl chloride and high-performance liquid chromatography coupled with Q-time-of-flight mass spectrometry. Talanta. 2011 Jan 15;83(3):751-6. doi: 10.1016/j.talanta.2010.10.039. Epub 2010 Nov 11. PMID 21147316
- [Background] Ivanova A, Qaqish BF, Schell MJ. Continuous toxicity monitoring in phase II trials in oncology. Biometrics. 2005 Jun;61(2):540-5. doi: 10.1111/j.1541-0420.2005.00311.x. PMID 16011702
- [Background] McCann PP, Pegg AE. Ornithine decarboxylase as an enzyme target for therapy. Pharmacol Ther. 1992;54(2):195-215. doi: 10.1016/0163-7258(92)90032-u. PMID 1438532